CLINICAL TRIAL: NCT05861297
Title: The Outcomes and Safety of Immunomodulators and Thrombopoietin Receptor Agonists in Primary Immune Thrombocytopenia Egyptian Patients With Hemorrhage Comorbidity
Brief Title: Immune Thrombocytopenia Management in Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nahda University (Other)
Responsible Party: Principal Investigator, Eman Mostafa Hamed, Teaching Assistant clinical pharmacy department, faculty of pharmacy, Nahda University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NahdaV
Record Dates: First submitted 2023-04-27; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Immune Thrombocytopenia Purpura
Keywords: Primary Immune Thrombocytopenia; Etrombopag; Dexamethasone; Romiplostim; Rituximab; Autoimmune Disorder
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Autoimmune Diseases | interventions — Dexamethasone; Prednisolone; Azathioprine; Rituximab; eltrombopag; romiplostim

STUDY DESIGN:
Intervention Model Description: comparsion between five groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Control group (Active Comparator): The first (control )group includes patients with confirmed diagnosed who received IV pulse (High Dose-Dexamethasone) therapy
  Interventions: Drug: Dexamethasone
- PSL - AZA group (Experimental): The second group includes patients with confirmed diagnosed who received Prednisolone -Azathioprine therapy
  Interventions: Drug: Prednisolone and Azathioprine
- The RTX group (Experimental): The third group includes patients with confirmed diagnosed who received Prednisolone -Azathioprine therapy
  Interventions: Drug: Rituximab
- The ELTRO group (Experimental): The fourth group includes patients with confirmed diagnosed who received E therapy
  Interventions: Drug: Eltrombopag
- The ROMP group (Experimental): The fifth group includes patients with confirmed diagnosed who received Romiplostim therapy
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Dexamethasone — Patients were initiated with High Dose-Dexamethasone with a dose of 40 mg/m2 daily for four days per week immediately after the diagnosis of ITP for 6 months
  Arms: Control group
Drug: Prednisolone and Azathioprine — the second group received 20 mg of Prednisolone three times daily and 1 mg/kg of oral Azathioprine once daily for two weeks, then tapering the Prednisolone dose through the subsequent weeks (6 weeks). While continuing treatment with Azathioprine for a total of six months.
  Arms: PSL - AZA group
Drug: Rituximab — The third group received 500 mg/m2 intravenously of Rituximab once weekly for one month
  Arms: The RTX group
Drug: Eltrombopag — The fourth group received 50 mg of Eltrombopag four hours before or after meals as oral daily doses for 6 months
  Arms: The ELTRO group
Drug: Romiplostim — The fifth group received 3μg/kg subcutaneous injection of Romiplostim once a week for 6 months
  Arms: The ROMP group

SUMMARY:
Immune thrombocytopenia treatment has evolved recently. However, none of treatments have only benefits without drawbacks. This study compares the clinical outcomes and adverse drug patterns of different treatment options. Medications which will be assessed during the current study are High Dose-dexamethasone (HD-DXM) (control group), Prednisolone + Azathioprine, Rituximab, Eltrombopag, and Romiplostim.

DETAILED DESCRIPTION:
A prospective controlled randomized study was conducted on primary Immune thrombocytopenia patients. The study's main objective is to evaluate the efficacy and adverse events profile of the different therapeutic approaches during Immune thrombocytopenia. Upon the confirmation of the Immune thrombocytopenia diagnosis, all patients immediately initiated the High Dose-dexamethasone as a frontline therapy for Immune thrombocytopenia with a dose of 40 mg/m2 daily for 4 days/week in the first month for one cycle. Then, the recruited patients who fulfilled the inclusion criteria are randomly assigned into one of five groups. Among these patients, the control group received IV pulse (HD-DXM) therapy with 40 mg/m2 daily for 4 successive days in a 28-day cycle to complete the six cycles. The Prednisolone + Azathioprine group received 20 mg of Prednisolone three times daily and 1 mg/kg of oral Azathioprine once daily for two weeks, then tapering the Prednisolone dose through the subsequent weeks (6 weeks). While continuing treatment with Azathioprine for a total of six months. The Rituximab group received 500 mg/m2 intravenously of Rituximab once weekly for one month. The Eltrombopag group received 50 mg of Eltrombopag four hours before or after meals as oral daily doses for 6 months. The Romiplostim group received 3μg/kg sub-cutaneous injection of Romiplostim once a week for 6 months. The first evaluation date of confirmed ITP diagnosis was well-defined as the first index date (baseline). After that, every patient visited the investigational site as the protocol prescribes once weekly to assess and adjust the doses of study medications. The outcome measures were judged at baseline, at the end of treatment (6 months), and after an additional 6-month free treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were adult patients aged 18 years or older, diagnosed with primary ITP after excluding secondary causes and with an initial PLTs count of less than 30 ×109/L or with hemorrhage manifestations.

Exclusion Criteria:

* Patients with a confirmed secondary ITP diagnoses such as (chemicals induced, systemic lupus erythematosus, immune thyroid diseases, a lymphoproliferative disease, or chronic infection, such as Helicobacter pylori, human immunodeficiency virus (HIV) or hepatitis C virus (HCV); with cardiac, renal, or liver disease; who had received NSAIDs or anti-platelets within one month before the initiation of the enrollment were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2024-01-18 (Estimated); Study Completion 2024-04-02 (Estimated)

PRIMARY OUTCOMES:
total patients who achieved sustained and overall response | 18 months
  The primary outcomes were the total percentage of patients achieving a sustained response (SR) till the end of the study, complete response (CR), and partial response (PR). CR was characterized by the absence of bleeding and an increase in the platelet count to above 100×109/L after one month of the treatment. SR was defined as achieving CR or partial response (PR) until the end of the study with a 2-fold upsurge from starting point [20, 21]. PR was represented as PLTs count ≥ 30×109/L after one month following therapy, and no response (NR) was defined as platelets < 30×109/L or bleeding

SECONDARY OUTCOMES:
number of patients relapsed and adverse events | 18 months
  The secondary outcome measures were a number of patients relapsed and adverse events (AEs). Relapse was pointed out as PLTs count below 30×109/L or bleeding episodes owing to thrombocytopenia afterward achieving the CR

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hussein Meabed, professor, Study Chair — faculty of medicine beni-suef university
Locations (1):
- EL-Kasr elineiy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamed EM, Ibrahim ARN, Meabed MH, Khalaf AM, El Demerdash DM, Elgendy MO, Saeed H, Salem HF, Rabea H. Therapeutic Outcomes of High Dose-Dexamethasone versus Prednisolone + Azathioprine, Rituximab, Eltrombopag, and Romiplostim Strategies in Persistent, Chronic, Refractory, and Relapsed Immune Thrombocytopenia Patients. Pharmaceuticals (Basel). 2023 Aug 29;16(9):1215. doi: 10.3390/ph16091215. PMID 37765023